CLINICAL TRIAL: NCT07066267
Title: Clinical Application of Autologous Adipose Stem Mitochondria Transplantation to Oocytes for Improving Embryo Quality in Patients With Recurrent Pregnancy Failure
Brief Title: Adipose Stem Cell Mitochondria Supplementation to Oocytes (ASCENT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunkaky Medical Cooperation (Industry)
Collaborators: Wish Fertility Hospital Pvt. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WishREC/24-011
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Female Infertility; Oocyte Competence; Mitochondria; Recurent Implantation Failures; Advanced Age
Keywords: mitochondria; mitochondria transplantation; Adipose stem cell; oocyte; Female infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: This is a triple-blind (Patient, Embryologist, Doctor), single-center, randomized, controlled experimental pilot study.
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Mitochondria transfer (Active Comparator): Mitochondria isolated from autologous adipose-derived stem cells are transplanted into the oocyte in conjunction with intracytoplasmic sperm injection (ICSI); Mito-ICSI group
  Interventions: Other: Experimental
- Conventonal Intracytoplasmic Sperm Injection (No Intervention): Conventional ICSI; Control group

INTERVENTIONS:
Other: Experimental — Autologous adipose stem cell mitochondrial transfer to mature oocytes along with intracytoplasmic sperm injection (ICSI). The intervention is also termed as Adipose Stem Cell ENergy Transfer (ASCENT).
  Arms: Autologous Mitochondria transfer

SUMMARY:
The purpose of this study is to investigate the potential of autologous adipose stem cell (ASC) mitochondrial transfer (ASCENT) to oocytes along with intracytoplasmic sperm injection (ICSI)as a means of enhancing embryo development and improving the success rate of in patients with a history of multiple IVF failures. Embryo quality plays a crucial role in determining the success of assisted reproductive technologies and directly contributes to repeated pregnancy failures. Several factors, including age, physiological conditions, genetics, and environmental influences, can significantly impact embryo quality. Oocytes, the largest cells in the human body, are heavily reliant on mitochondria. Mitochondria's role in providing energy for oocytes is crucial, and insufficient energy production has been linked to poor oocyte and embryo quality. Some human studies have shown that increasing oocyte mitochondrial mass can improve embryo quality in patients who have experienced repeated IVF failures.

DETAILED DESCRIPTION:
Sibling mature oocytes will be randomly divided into two groups. And one group of oocytes will be undergone conventional intracytoplasmic sperm injection (ICSI) (control group; cont. ICSI) and the other group of oocytes will be undergone mitochondria transplantation along with intracytoplasmic sperm injection (Mito-ICSI). Viable blastocysts from both groups will be biopsied for preimplantation genetic testing for aneuploidy.

ELIGIBILITY:
Inclusion Criteria:

* Having at least three previous failed IVF trial
* Specifically consented for to collect biopsies for Preimplantation generic testing for aneuploidy (PGTA) analysis
* Specifically consented for to have single blastocyst transfer (recommended)
* No major uterine or ovarian abnormalities
* Specifically consented for to have all embryos frozen
* Specifically consented for to collect adipose tissues from subcutaneous liposuction
* BMI level level <26kg/m2

Exclusion Criteria:

* Ovarian endometriosis with Chocolate cysts (American Fertility Society (AFS)) classification type 3 and 4
* Any medical contraindication oocyte retrieval or subsequent procedures Ovarian hyperstimulation syndrome Bleeding disorders Sex hormone allergies Severe emotional defect on injections
* Severe sperm abnormalities
* <5 million/mL motile sperm
* Uterine structural anomalies
* Polycystic ovaries
* Premature ovarian failure

Ages: 29 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Embryo development rate | Up to 8 weeks post-intervention
  Analyze and compare the transferable embryo rate per zygote on day 3 & day 5 between the Intervention and control groups.

SECONDARY OUTCOMES:
Ongoing clinical pregnancy rate after the first transfer | Up to 18 months post-intervention
  Compare ongoing clinical pregnancy rates between the intervention and conrolgroups
Chemical pregnancy rate | Up to 18 months post-intervention
  Compare the chemical pregnancy rates between the two groups.
Live Birth rates | Up to 24 months post-intervention
  Compare live Birth rate following the intervention in both groups
Pregnancy complication | Up to 24 months post-intervention
  Rate of pregnancy complication in both groups
Abortion rate | Up to 24 months post-intervention
  Compare the abortion rates in both groups
Additional in vitro fertilization - outcome indicators | Up to 8 weeks post-intervention
  Compare the rate of fertilization in between two groups
Additional in vitro fertilization - outcome indicators | Up to 8 weeks post-intervention
  Rate of abnormal fertilization in both groups
Additional in vitro fertilization - outcome indicators | Up to 8 weeks post-intervention
  The rate of non-transferable embryos in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Helaruwan Pasan Kumara WA, MD, PhD, Principal Investigator — Wish Fertility Hospital Pvt. Ltd; Prof. Yoshiharu Morimoto, MD, PhD, Principal Investigator — Horac Grand Front Osaka Clinic
Locations (1):
- Wish Fertility Hospital Pvt. Ltd, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Result] Kankanam Gamage US, Hashimoto S, Miyamoto Y, Nakano T, Yamanaka M, Koike A, Satoh M, Morimoto Y. Mitochondria Transfer from Adipose Stem Cells Improves the Developmental Potential of Cryopreserved Oocytes. Biomolecules. 2022 Jul 21;12(7):1008. doi: 10.3390/biom12071008. PMID 35883564
- [Result] Kankanam Gamage SU, Hashimoto S, Miyamoto Y, Nakano T, Yamanaka M, Kitaji H, Takada Y, Matsumoto H, Koike A, Satoh M, Ichishi M, Watanabe M, Morimoto Y. Supplementation with autologous adipose stem cell-derived mitochondria can be a safe and promising strategy for improving oocyte quality. J Assist Reprod Genet. 2024 Aug;41(8):2065-2077. doi: 10.1007/s10815-024-03137-2. Epub 2024 May 22. PMID 38777961
- [Result] Morimoto Y, Gamage USK, Yamochi T, Saeki N, Morimoto N, Yamanaka M, Koike A, Miyamoto Y, Tanaka K, Fukuda A, Hashimoto S, Yanagimachi R. Mitochondrial Transfer into Human Oocytes Improved Embryo Quality and Clinical Outcomes in Recurrent Pregnancy Failure Cases. Int J Mol Sci. 2023 Feb 1;24(3):2738. doi: 10.3390/ijms24032738. PMID 36769061